CLINICAL TRIAL: NCT00002449
Title: A Bridging Dose-Escalation Study of the Safety, Pharmacokinetic Properties, and Immunologic Effect of Subcutaneous L2-7001 (Recombinant Human Interleukin-2) in Patients Infected With HIV With CD4+ T-Cell Counts of 300 to 500 Cells/mm3 and Viral Burden Under 10,000 Copies/Ml on Active Antiretroviral Therapy (ART)
Brief Title: Safety and Effectiveness of L2-7001 (Interleukin-2) in HIV-Positive Patients Receiving Anti-HIV Therapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chiron Corporation (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: B007; CS-MM-9901
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-07

CONDITIONS: HIV Infections
Keywords: Recombinant Proteins; Injections, Subcutaneous; Interleukin-2; Dose-Response Relationship, Drug; CD4 Lymphocyte Count; Anti-HIV Agents; Viral Load; Pharmacokinetics
MeSH Terms: conditions — HIV Infections | interventions — aldesleukin

INTERVENTIONS:
Drug: Aldesleukin

SUMMARY:
The purpose of this study is to see if it is safe and effective to give HIV-positive patients L2-7001 (a type of interleukin-2) plus anti-HIV therapy. Interleukin-2 (IL-2) is a substance naturally produced by the body's white blood cells that plays an important role in helping the body fight infection. IL-2 may be able to boost the immune systems of people with HIV infection.

DETAILED DESCRIPTION:
This study takes place in two phases. Phase A consists of an open-label dose-escalation of L2-7001 through four dose levels. Ascending dose cohorts of five patients are studied. The safety and tolerability of L2-7001 is assessed in preparation for the second phase of the study and to estimate an MTD. Phase B involves randomization of 190 patients to (a) one of three dose levels of L2-7001 plus ART, (b) one of two dosing levels of Proleukin plus ART, or (c) ART alone. L2-7001 and Proleukin are given SC every 12 hours for the first 5 days of an 8-week cycle for three cycles. Serum IL-2 levels, soluble IL-2 receptor levels, and levels of pro-inflammatory cytokines are evaluated in 8 patients randomized to each treatment cohort of Phase B. All patients completing this phase of the protocol are eligible to be screened for enrollment in a maintenance use protocol which will allow for access to L2-7001.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have a viral load below 10,000 copies/ml.
* Have a CD4 count between 300 and 500 cells/mm3.
* Have been on stable anti-HIV therapy for 4 months. Patients must be taking at least 2 drugs, 1 of which must be a protease inhibitor or a nonnucleoside drug (NNRTI).
* Are at least 18 years old.
* Agree to use an effective barrier method of birth control, such as condoms, during the study.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have an AIDS-defining illness. (Patients who have had an AIDS-defining illness that was cured may still be eligible.)
* Have an alcohol or drug abuse problem that the doctors feel would affect their ability to participate.
* Have cancer requiring chemotherapy.
* Have a history of autoimmune disease.
* Have uncontrolled diabetes or certain thyroid problems.
* Have mental illness or other serious medical condition that the doctors feel would affect their ability to participate.
* Have received IL-2 in the past.
* Have taken corticosteroids or certain medications that affect the immune system in the past 4 weeks.
* Have taken hydroxyurea in the past 4 months.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212
Dates: Start 1999-08

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Sorra Research Ctr / Med Forum, Birmingham, Alabama
  - Pacific Oaks Research, Beverly Hills, California
  - Orange County Ctr for Special Immunology, Fountain Valley, California
  - St Lukes Medical Group, San Diego, California
  - Kaiser Foundation Hospital, San Francisco, California
  - Denver Inf Disease Consultants, Denver, Colorado
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - Community AIDS Resource Inc, Coral Gables, Florida
  - Steinhart Medical Associates, Miami, Florida
  - Specialty Med Care Ctrs of South Florida Inc, Miami, Florida
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Northstar Med Clinic, Chicago, Illinois
  - Fenway Community Health Ctr, Boston, Massachusetts
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Albany Med College, Albany, New York
  - Anderson Clinical Research Inc, Rego Park, New York
  - Associates in Med and Mental Health, Tulsa, Oklahoma
  - Research and Education Group, Portland, Oregon
  - Anderson Clinical Research, Pittsburgh, Pennsylvania
  - Central Texas Clinical Research, Austin, Texas
  - N Texas Ctr for AIDS & Clin Rsch, Dallas, Texas
  - Gathe, Joseph, M.D., Houston, Texas
  - Virginia Mason Med Ctr, Seattle, Washington